CLINICAL TRIAL: NCT03155425
Title: An Open-Label, Single Arm, Multi-Center, Phase 2 Study of PD-1 Antibody SHR-1210 in Subjects With Relapsed or Refractory Classic Hodgkin's Lymphoma
Brief Title: PD-1 Antibody SHR-1210 in Patients With Relapsed or Refractory Classic Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-204
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-04

CONDITIONS: Hodgkin Lymphoma, Adult
MeSH Terms: conditions — Hodgkin Disease | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection SHR-1210 (Experimental): SHR-1210 injection, 200 mg/dose, intravenous infusion.
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — A humanized monoclonal immunoglobulin

SUMMARY:
This is an open-label, multicenter, non-randomized, phase 2 trial to evaluate efficacy and safety of SHR-1210 in patients with relapsed or refractory classic Hodgkin's lymphoma. The primary objective is to assess ORR of SHR-1210 in patients with relapsed or refractory classic Hodgkin's lymphoma.

DETAILED DESCRIPTION:
The primary objective of this phase 2 study is to assess objective response rate of SHR-1210 in patients with relapsed or refractory classic Hodgkin's lymphoma. The secondary objective is to observe the duration of response, progression free survival, time to response, overall survival and safety of SHR-1210 in relapsed or refractory classic Hodgkin's lymphoma. Pharmacokinetic index is also investigated in 12 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed classic Hodgkin's lymphoma;
2. Relapsed or refractory cHL and meet any of the following criterions: a) did not achieve remission or progression after autologous hematopoietic stem cell transplantation. b) at least 2 lines of systemic chemotherapy and are not suitable for autologous stem cell transplantation;
3. Subjects enrolled have measurable lesion (s) according to Lugano 2014 criteria;
4. ECOG performance status of 0 or 1;
5. Life expectancy ≥ 12 weeks;
6. Adequate laboratory parameters during the screening period as evidenced by the following:

   1. Absolute neutrophil count ≥ 1.0 × 109/L;
   2. Platelets ≥ 75 × 109/L;
   3. Hemoglobin ≥ 8.0 g/dL;
   4. Total bilirubin (TBIL) < 1.5 × upper limit of normal (ULN), ALT and AST ≤ 2.5×ULN;
   5. Serum Creatinine ≤1.25×ULN or Creatinine clearance≥45 mL/min;
   6. Coagulation function index: INR ≤1.5×ULN，APTT≤1.5×ULN;
7. Women of childbearing potential (WOCBP) must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 60 days after receiving the last dose of study treatment. Women of childbearing potential with pregnancy test negative within 7 days before entering the group; male subjects with WOCBP partner should receive Surgical sterilization or consent to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 120 days after receiving the last dose of study treatment;
8. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Known nodular lymphoma predominant Hodgkin lymphoma or Grey zone lymphoma.
2. Known central nervous system lymphoma.
3. History and complication:

(1) Active, known or suspected autoimmune disease. Subjects who were in a stable state without systemic immunosuppressive therapy were admitted; (2) Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic corticosteroids > 10mg; doses > 10 mg/day topical prednisone or equivalent are prohibited within 2 weeks before entering the group; (3) Received anti-tumor vaccines or other anti-tumor therapy with immune stimulation within 3 months before the first dose SHR-1210; (4) Prior exposure to any PD-1/PD-L1/PD -L 2 or CTLA -4 antibody; (5) Participating in other clinical studies or less than 4 weeks before the end of a clinical trial; (6) Known and highly Suspicion of interstitial pneumonia; (7) Other active malignancies that required treating. (subjects with skin basal cell carcinoma, superficial bladder cancer, skin squamous cell carcinoma or cervical carcinoma who had no disease recurrence within 5 years after the start of treatment were excluded); (8) Received chemotherapy, radiotherapy, immunotherapy, including topical therapy within 4 weeks. Previous anti-tumor therapy related adverse reactions (except hair loss) did not recover to CTCAE ≤1; (9) Prior allo-HSCT; (10) ASCT within 90 days; (11) Impact of major surgery or severe trauma had been eliminated for less than 14 days; (12) Active pulmonary tuberculosis; (13) Severe acute or chronic infection requiring systemic therapy; (14) Suffering from heart failure (New York Heart Association standard III and given appropriate medical treatment. Uncontrolled coronary artery disease and arrhythmia. History of myocardial infarction within 6 months; (15) Inoculated with live vaccine within 4 weeks before receiving the investigational drug. Injections of inactivated influenza vaccine for seasonal influenza are permitted, but not live attenuated influenza vaccines for intranasal use.

4. laboratory test:

(1) known HIV positive or known AIDS; (2) Untreated active hepatitis; co-infection with hepatitis B and hepatitis C.

5. Other factors that may lead to the study termination, such as severe disease or abnormal laboratory tests or family or social factors affecting subjects safety or test data and sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Xiao, MD, Study Director — Jiangsu Hengrui Pharmaceutical Co., Ltd.
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Song Y, Wu J, Chen X, Lin T, Cao J, Liu Y, Zhao Y, Jin J, Huang H, Hu J, Luo J, Zhang L, Xue H, Zhang Q, Wang W, Chen C, Feng J, Zhu J. A Single-Arm, Multicenter, Phase II Study of Camrelizumab in Relapsed or Refractory Classical Hodgkin Lymphoma. Clin Cancer Res. 2019 Dec 15;25(24):7363-7369. doi: 10.1158/1078-0432.CCR-19-1680. Epub 2019 Aug 16. PMID 31420358

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Injection SHR-1210
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Injection SHR-1210
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 34 [20 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 75
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 75

OUTCOME MEASURES:

1. Primary Outcome: ORR Assess by IRC
Description: rate of subjects achieved complete response plus partial response in all evaluable subjects (Response was assessed with CT and PET using 2014 Lugano Criteria for Malignant Lymphomas, CR is disappearance of all tumor lesions, PR is over 50% decrease of the sum of the product of the perpendicular diameters from baseline ;overall response:PR+CR)
Time Frame: CT was conducted at baseline, at weeks 9, 17, 25, 37, 49, 65, 81, and 97, and then every 26 weeks; PET was conducted at baseline, weeks 17 and 25. ORR of 36 weeks based on CT and PET were reported.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Injection SHR-1210
Number analyzed (Participants) | 75
percentage | 76.0 [64.7 to 85.1]

2. Secondary Outcome: DoR Assess by IRC
Description: Duration of Response (Response was assessed with CT and PET using 2014 Lugano Criteria for Malignant Lymphomas, disease progression is over 50% increase of an product of perpendicular diameters of any target lesion from nadir with any diameter increased over 0.5cm for lesions <=2cm or increased by 1cm for lesions >2cm，or appearance of new lesions, or progression of non-target lesion )
Time Frame: CT was conducted at baseline, at weeks 9, 17, 25, 37, 49, 65, 81, and 97, and then every 26 weeks; PET was conducted at baseline, weeks 17 and 25. DoR of 36 weeks based on CT and PET were reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Injection SHR-1210
Number analyzed (Participants) | 75
months | 31.7 [16.7 to NA] — insufficient number of patients with events

3. Secondary Outcome: PFS Assess by IRC
Description: Progression-free Survival (Response was assessed with CT and PET using 2014 Lugano Criteria for Malignant Lymphomas, disease progression is over 50% increase of an product of perpendicular diameters of any target lesion from nadir with any diameter increased over 0.5cm for lesions <=2cm or increased by 1cm for lesions >2cm，or appearance of new lesions, or progression of non-target lesion )
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Injection SHR-1210
Number analyzed (Participants) | 75
months | 22.5 [14.7 to NA] — insufficient number of patients with events

4. Secondary Outcome: TTR Assess by IRC
Description: Time to response (Response was assessed with CT and PET using 2014 Lugano Criteria for Malignant Lymphomas, CR is disappearance of all tumor lesions, PR is over 50% decrease of the sum of the product of the perpendicular diameters from baseline ;overall response:PR+CR)
Time Frame: CT was conducted at baseline, at weeks 9, 17, 25, 37, 49, 65, 81, and 97, and then every 26 weeks; PET was conducted at baseline, weeks 17 and 25.
Measure: Median (Full Range); unit: months
Arm/Group | Injection SHR-1210
Number analyzed (Participants) | 75
months | 2.0 [1.7 to 5.7]

5. Secondary Outcome: OS
Description: Overall Survival
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Injection SHR-1210
Number analyzed (Participants) | 75
months | NA [NA to NA] — insufficient number of patients with events

6. Secondary Outcome: Incidence and Severity of Adverse Events (AE)
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Injection SHR-1210
Number analyzed (Participants) | 75
participants | 75

ADVERSE EVENTS:
Time Frame: 3 years
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Injection SHR-1210
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 12/75
Other Adverse Events (participants affected / at risk) | 74/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Injection SHR-1210 (N=75)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Immune-Mediated Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Soft Tissue Infection (Infections and infestations) | 1
Blood Bilirubin Increased (Investigations) | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1
Chest Discomfort (General disorders) | 1
Inflammation (General disorders) | 1
Tumor Pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Immune System Disorders (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nasal Mucosa Reactive Capillary Endothelial Proliferation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Reactive Cutaneous Capillary Endothelial Proliferation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nephrotic Syndrome (Renal and urinary disorders) | 1
Renal Injury (Renal and urinary disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Injection SHR-1210 (N=75)
Anaemia (Blood and lymphatic system disorders) | 17
Arrhythmia (Cardiac disorders) | 4
Hypothyroidism (Endocrine disorders) | 24
Hyperthyroidism (Endocrine disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 8
Pyrexia (General disorders) | 33
Asthenia (General disorders) | 6
Reactive angioendotheliomatosis (Immune system disorders) | 73
Upper respiratory tract infection (Infections and infestations) | 41
Nasopharyngitis (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 9
Herpes zoster (Infections and infestations) | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 12
Alanine aminotransferase increased (Investigations) | 22
White blood cell count decreased (Investigations) | 22
Neutrophil count decreased (Investigations) | 19
Weight increased (Investigations) | 19
Aspartate aminotransferase increased (Investigations) | 17
Blood thyroid stimulating hormone increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 12
Platelet count decreased (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 11
Lymphocyte count decreased (Investigations) | 7
Protein urine present (Investigations) | 7
Weight decreased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 6
Electrocardiogram QT prolonged (Investigations) | 6
Bilirubin conjugated increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 5
Blood uric acid increased (Investigations) | 5
Blood bilirubin unconjugated increased (Investigations) | 4
Blood glucose increased (Investigations) | 4
Occult blood positive (Investigations) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hyperuricaemia (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 4
Proteinuria (Renal and urinary disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03155425/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT03155425/SAP_001.pdf